CLINICAL TRIAL: NCT01600898
Title: Screening and Risk Factors of Pulmonary Arterial Hypertension in BMPR2 Mutation Asymptomatic Carriers
Brief Title: Screening of Pulmonary Arterial Hypertension in BMPR2 Mutation Carriers
Acronym: DELPHI-2
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P100104; AOM 10175 (Other: PHRC 2010)
Record Dates: First submitted 2012-05-15; First posted 2012-05-17 (Estimated); Last update posted 2021-01-13 (Actual); Status verified 2019-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Asymptomatic carriers of a BMPR2 mutation; follow up study
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Asymptomatic BMPR2 mutation carriers: Asymptomatic BMPR2 mutation carriers

SUMMARY:
In this prospective study, the investigators will implement a systematic screening program and 3-year follow-up in a cohort of asymptomatic BMPR2 mutation carriers. This study is designed to:

* determine predictive factors (biological, functional, radiological and hemodynamic) of development of PAH
* monitor these subjects' clinical, functional, biological, echocardiographic and hemodynamic characteristics
* assess the risk of occurrence of PAH
* screen patients with PAH at an early stage of disease and offer them an early management
* constitute a collection of biological samples (0, 12, 24 months follow-up) of asymptomatic BMPR2 mutation carriers.

DETAILED DESCRIPTION:
Introduction:

Pulmonary arterial hypertension is characterized by remodeling of small pulmonary arteries leading to a progressive increase in pulmonary vascular resistance resulting to right heart failure and ultimately death. The disease is diagnosed when symptomatic, demonstrating the existence of an already advanced form of the disease. Indeed, there is no simple tool allowing an early diagnosis of PAH and the disease is usually diagnosed in advanced stages. Diagnostic confirmation of PAH is based on the elevation of mean pulmonary arterial pressures measured during right heart catheterization. Despite the development of specific treatment in recent years, PAH remains a disease with poor prognosis, for which no cure is possible, apart from lung transplantation in selected cases. However recent studies have shown that specific drug therapy in early disease stages could improve the prognosis of this life threatening disease. This is why it seems important to establish early diagnosis of PAH, especially in high-risk populations such as asymptomatic carriers of BMPR2 (Bone Morphogenetic Protein Receptor 2) mutations. PAH due to BMPR2 mutations is an autosomal dominant disease with incomplete penetrance. Even if there are no accurate data in the literature, it is estimated that 20% of patients with BMPR2 mutations develop PAH in the course of their life. The implementation of a genetic counseling in the National Reference Center for Severe Pulmonary Hypertension (BICETRE Hospital) allowed us to propose systematic assessment of BMPR2 mutations in patients with idiopathic or familial PAH. In 2012 we identified 130 PAH patients carriers of a BMPR2 mutation. This approach has enabled the detection of families at risk for PAH and to offer genetic counseling to the asymptomatic relatives with BMPR2 mutation. However, data on the evolution of asymptomatic carriers of BMPR2 mutation are lacking. Furthermore, there is no available consensus or guideline on how to follow this population. To date, it is not possible to differentiate asymptomatic subjects carrying BMPR2 mutations that will develop PAH from those who will never develop this disease. However, given the high risk of these subjects to develop PAH (risk of 20% against 25/million in the general population), and the limited knowledge of characteristics of this population, it seems essential to offer a prospective follow-up to this population at risk.

Aim and objective:

The main objective of this study to is follow prospectively for 3 years a cohort of asymptomatic carriers of BMPR2 mutation to:

* determine predictive factors (biological, functional, radiological and hemodynamic) of development of PAH
* monitor these subjects' clinical, functional, biological, echocardiographic and hemodynamic characteristics
* assess the risk of occurrence of PAH
* screen patients with PAH at an early stage of disease and offer them an early management
* constitute a collection of biological samples (0, 12, 24 months follow-up) of asymptomatic BMPR2 mutation carriers.

Methodology :

Evaluation of subjects at inclusion after informed consent (Ethics Committee approval obtained since 2011):

* Clinical evaluation: dyspnea assessed by NYHA functional class (I-IV), signs of right heart failure
* Chest radiograph, electrocardiogram
* Right heart catheterization (in a subset of volunteers): measurement of mean pulmonary artery pressure, pulmonary artery occlusion pressure (PAOP) and cardiac output (CO) at rest and during exercise
* Echocardiography: measurement of the velocity of tricuspid regurgitation (VIT), measurement of TAPSE and Tei index, pericardial effusion, dilatation and hypertrophy of the right ventricle
* Stress Test: VO2 peak and VO2 specific, VE minute ventilation, VD / VT dead space, ventilatory reserve, alveolar-arterial gradient, pulse oxygen, PaO2
* Lung function tests: measurement of DLCO and DLNO
* Magnetic resonance imaging (MRI) measuring end systolic diastolic volumes of the right ventricle, right ventricular mass, septal curvature, diameter of the pulmonary arteries, surface of the right atrium
* Biology: Determination of plasma NT-proBNP, uric acid, serum sodium, creatinine, PDGF, ET-1, ET-3, CRPus, IL-6, soluble c-kit, CXCL12, progenitors and circulating fibrocytes

Subjects will be evaluated as outpatients scheduled to the National Reference Center for Severe Pulmonary Hypertension 12, 24 and 36 months after inclusion or if symptoms appear (dyspnoea, right heart failure, malaise or syncope).

During these consultations, the assessment will include: clinical evaluation, chest radiograph, electrocardiogram, echocardiogram, stress testing, pulmonary function tests, magnetic resonance imaging, and biology.

To confirm the suspicion of PAH and assess their severity, right heart catheterization at rest and during exercise will be offered according to a decision algorithm.

Right heart catheterization will be performed if one of the following abnormalities is found:

* Dyspnea, malaise or unexplained syncope
* Tricuspid regurgitation velocity ≥ 2.8 m / s
* Decrease of the specific peak VO2 ≥ 20% as compared to the gold standard

If diagnosis of PAH is confirmed, patients will be treated according to the recently updated recommendations of the European Respiratory Society and European Society of Cardiology.

ELIGIBILITY:
Inclusion Criteria:

* men and women over 18 years old,
* carriers of a BMPR2 mutation without known PAH,
* having given his informed consent

Exclusion Criteria:

* men and women under 18 years old,
* patients with a known PAH,
* pregnant women,
* adults protected,
* detainees,
* people in emergencies,
* people refusing or unable to give informed consent,
* no affiliation to a regime of social security.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: asymptomatic BMPR2 mutation carriers.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2012-03; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
predictive factors of the occurrence of PAH | 2 years
  follow prospectively a cohort of asymptomatic BMPR2 mutation carriers to determine predictive factors of the occurrence of PAH.

SECONDARY OUTCOMES:
Evolution of characteristics of asymptomatic BMPR2 mutation carriers | 2 years
  monitor these subjects' clinical, functional, biological, echocardiographic and hemodynamic characteristics, assess the risk of occurrence of PAH , screen patients with PAH at an early stage of disease and offer them an early management, constitute a collection of biological samples (0, 12, 24 months follow-up) of asymptomatic BMPR2 mutation carriers.

CONTACTS AND LOCATIONS:
Overall Officials: David Montani, Md, PhD, Principal Investigator — Assistance-Publique Hôpitaux de Paris, Hôpital Bicêtre, Service de pneumologie
Locations (1):
- David Montani, Le Kremlin-Bicêtre, France

REFERENCES:
- [Result] Montani D, Girerd B, Jais X, Laveneziana P, Lau EMT, Bouchachi A, Hascoet S, Gunther S, Godinas L, Parent F, Guignabert C, Beurnier A, Chemla D, Herve P, Eyries M, Soubrier F, Simonneau G, Sitbon O, Savale L, Humbert M. Screening for pulmonary arterial hypertension in adults carrying a BMPR2 mutation. Eur Respir J. 2021 Jul 22;58(1):2004229. doi: 10.1183/13993003.04229-2020. Print 2021 Jul. PMID 33380512
- See also: We thank the funding program PHRC that funded this study. We thank the Clinical Research Unit Paris Sud (Bicetre hospital - APHP) for monitoring and coordinating this study. — http://hopitaux-paris-sud.aphp.fr/la-recherche-medicale-du-groupe-hospitalier-3/les-structures-de-la-recherche/